CLINICAL TRIAL: NCT05943353
Title: The Efficacy of Pentoxifylline on Sperm Selecting in Intracytoplasmic Sperm Injection (ICSI) of Absolute Asthenozoospermia
Brief Title: ICSI Using Pentoxifylline to Identify Viable Spermatozoa in Absolute Asthenozoospermia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 07/23/DD-BVMD
Record Dates: First submitted 2023-07-03; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: in Vitro Fertilization
Keywords: Pentoxifylline; Sperm selecting; Absolute asthenozoospermia; in Vitro Fertilization
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- non-randomized trials (Other)
  Interventions: Other: Pentoxifylline

INTERVENTIONS:
Other: Pentoxifylline — Prominently, Pentoxyfilline (PTX) is a methylxanthine derivative, is an inhibitor of phosphodiesterase activity and increases intracellular cAMP levels, which play an important role in sperm motility. The ability of PTX to improve sperm motility was first recognized in the study of Turner et al (1978). One of the advantages of PTX is that it significantly reduces the time to find and select motile sperm in cases of completely immotile sperm. In recent years, many studies have demonstrated the effectiveness of PTX for the group of spermatozoa, sperm carrying severe abnormalities. Therefore, the use of a sperm motility inducer such as PTX is a potential method to replace traditional ICSI sperm selection methods. Therefore, we performed this study with the aim to evaluate the effectiveness of PTX to select sperm in ICSI on the group of sperm that were completely immotile after ejaculation and obtained from the procedure.

SUMMARY:
Absolute asthenozoospermia is a rare condition in men with an occurrence frequency of 1/5000 and greatly affects fertility product. Previous studies have shown that the ovum can be fertilized with live but immotile sperm. However, the selection of live sperm for ICSI in immotile sperm samples is challenging for embryologists. Prominently, Pentoxyfilline (PTX) is a methylxanthine derivative, is an inhibitor of phosphodiesterase activity and increases intracellular cAMP levels, which play an important role in sperm motility. In recent years, many studies have demonstrated the effectiveness of PTX for the group of spermatozoa, sperm carrying severe abnormalities. In Vietnam, the application of PTX in ICSI has not yet been done in assisted reproductive centers. It is necessary to evaluate the effectiveness of PTX on ICSI treatment results in order to replace traditional methods and optimize treatment outcomes for patients.

DETAILED DESCRIPTION:
Sperm motility is an important factor in sperm selection for intracytoplasmic sperm injection. Intracytoplasmic Sperm Injection (ICSI), affects the success of ICSI cycles. In cases of severe male factor infertility, if motile sperm are still observed, ICSI still has the potential to help improve fertilization rates and treatment outcomes for patients. In contrast, the absence of motile sperm after ejaculation greatly affects the fertilization rate and the success of the ICSI cycle.

Absolute asthenozoospermia is a rare condition in men with an occurrence frequency of 1/5000 and greatly affects fertility product. In addition, complete immobility of sperm was also observed in cases of sperm collection from epididymal surgery (Percutaneous Epididymal Sperm Aspiration (PESA) or obtained from the testicles (Testicular Sperm Extraction (TESE). The characteristics of sperm samples obtained from the procedure are usually a high percentage of poor motility or complete immobility and cryopreservation of sperm may affect sperm motility and viability, especially for sperm samples from surgical collection.

Previous studies have shown that the ovum can be fertilized with live but immotile sperm. However, the selection of live sperm for ICSI in immotile sperm samples is challenging for embryologists. Currently, the methods performed in this case include the hypo-osmotic swelling test (HOS test), the sperm tail flexibility test (STFT) and laser-assisted immotile sperm selection (LAISS). However, traditional methods such as HOS test and STFT have the common disadvantage of long operation time and the result of sperm selection can be false positive, LAISS method is reported to be highly effective but still has some negative effects disadvantages in terms of operation time, high operating costs and requiring professional qualifications. Besides the above methods, the use of chemical inducers for sperm selection has received more and more attention in recent years. Prominently, Pentoxyfilline (PTX) is a methylxanthine derivative, is an inhibitor of phosphodiesterase activity and increases intracellular cAMP levels, which play an important role in sperm motility. The ability of PTX to improve sperm motility was first recognized in the study of Turner et al (1978). One of the advantages of PTX is that it significantly reduces the time to find and select motile sperm in cases of completely immotile sperm. In recent years, many studies have demonstrated the effectiveness of PTX for the group of spermatozoa, sperm carrying severe abnormalities. The study of Kovacic et al (2006) compared the embryology results of two groups of ICSI from spermatozoa with and without PTX use, in addition, the average ICSI time of 1 cycle (from time to time) initiation of sperm selection and immobilization until completion of the ICSI procedure) were evaluated in two groups. PTX shortened ICSI time (mean 30 minutes) compared with the control group (mean 120 minutes). In addition, when compared with the group that did not use PTX, the group that used PTX had higher fertilization results (66% vs 50.9%, P < 0.005) and a higher clinical pregnancy rate (38.3%) compared to 26.7%).

In addition, the use of PTX is assessed to have no negative impact on sperm and the health of live children. Stephanie et al (2021) evaluated the effects of PTX use on the development and behavior of 3-year-old children born from the ICSI cycle. No abnormal growth was observed among 8 children born from ICSI-PTX cycle compared with 6/170 children in the control group (0% vs 3.5%, P=0.28). In addition, there was no difference in the percentage of children with behavioral abnormalities in the ICSI-PTX group compared with the control group (0% vs. 9.4%, P=1.00). The study showed that PTX has potential applications in ICSI to improve sperm motility in cases of complete immobility, helping to improve treatment outcomes for patients. Therefore, the use of a sperm motility inducer such as PTX is a potential method to replace traditional ICSI sperm selection methods. In Vietnam, the application of PTX in ICSI has not yet been done in assisted reproductive centers. It is necessary to evaluate the effectiveness of PTX on ICSI treatment results in order to replace traditional methods and optimize treatment outcomes for patients. Therefore, the investigators performed this study with the aim to evaluate the effectiveness of PTX to select sperm in ICSI on the group of sperm that were completely immotile after ejaculation and obtained from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Sperm are completely immotile since PESA, TESE and MicroTESE
* Sperm are completely immotile after ejaculation

Exclusion Criteria:

* Oocyte maturation cycle in vitro

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | 16-18 hours after ICSI-PTX
  Total number of zygotes fertilized / total number of MII oocytes. zygote sperm is defined as a 2PN zygote at the time of testing fertilization17±1hours after ICSI

SECONDARY OUTCOMES:
Rate of good embryos on day 3 | 67-69 hours
  Total number of day 3 and type 2 embryos / total number of day 3 embryos at the time of embryo examination. Standard for grading embryo quality according to consensus Alpha and ESHRE (2011)
Rate of good embryos on day 5 | 114-118 hours
  Total number of day 5 embryos type 1 and type 2 / total number of day 3 embryos at the time of day 5 embryo examination. Standard for grading embryo quality according to consensus Alpha and ESHRE (2011)
Clinical pregnancy rate | Clinical pregnancy is defined as the presence of an intrauterine gestational sac on ultrasound from 5 weeks of age
  Calculated by the number of clinical pregnancies / total number of patients participating in the study.
Progressing pregnancy rate | An advanced pregnancy was defined as having at least one gestational sac with a fetal heartbeat up to 12 weeks of age
  Calculated by the number of active pregnancies/total number of patients participating in the study.
Miscarriage rate | Progressive miscarriage is defined as: before the end of the 22nd week of pregnancy in which the fetus is no longer viable and expelled from the uterus.
  Calculated by the number of cases of ongoing miscarriage / total number of patients participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, M.D, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- IVFMD, My Duc Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No